CLINICAL TRIAL: NCT04566016
Title: General Versus Regional Anaesthesia in Peripheral Arterial Surgery: Effects on the Incidence of Postoperative Pulmonary Complications.
Brief Title: General Versus Regional Anaesthesia in Peripheral Arterial Surgery: Incidence of Postoperative Pulmonary Complications.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 95165518.6.0000.5327; RBR-72fpz2 (Other: Registro Brasileiro de Ensaios Clínicos (ReBEC))
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Peripheral Vascular Diseases
Keywords: postoperative pulmonary complications; vascular surgery; regional anesthesia; mechanical ventilation
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Anesthesia, Conduction; Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: Randomized parallel controlled trial.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regional anesthesia (Experimental): Patients scheduled for lower limb arterial bypass surgery and allocated for treatment with spinal anesthesia associated with spontaneous ventilation (nasal cannula with supplemental oxygen - Group 1).
  Interventions: Procedure: Regional anesthesia
- General anesthesia (Active Comparator): Patients scheduled for lower limb arterial bypass surgery and allocated for treatment with general anesthesia under controlled mechanical ventilation (tidal volume 6 to 8 ml / kg of the predicted body weight and PEEP of 5 cmH2O - Group 2).
  Interventions: Procedure: Regional anesthesia

INTERVENTIONS:
Procedure: Regional anesthesia — Patients scheduled for lower limb arterial bypass surgery will be randomly allocated for treatment with spinal anesthesia associated with spontaneous ventilation (nasal cannula with supplemental oxygen - Group 1) or treatment with general anesthesia under controlled mechanical ventilation (tidal volume 6 to 8 ml / kg of the predicted body weight and PEEP of 5 cmH2O - Group 2).
  Other Names: Spinal anesthesia

SUMMARY:
The study will be designed as a prospective clinical trial. Patients scheduled for lower limb arterial bypass surgery will be randomly allocated for treatment with spinal anesthesia associated with spontaneous ventilation (nasal cannula with supplemental oxygen - Group 1) or treatment with general anesthesia under controlled mechanical ventilation (tidal volume 6 to 8 ml / kg of the predicted body weight and PEEP of 5 cmH2O - Group 2).

DETAILED DESCRIPTION:
In this prospective and randomized study, only adult ASA II to IV patients, aged over 18 years, scheduled to undergo lower limb arterial revascularization surgery at the Hospital de Clínicas in Porto Alegre and at the Hospital Nossa Senhora da Conceição will be included.

The study will be designed as a prospective clinical trial. Patients will be randomly allocated for treatment with spinal neuraxial anesthesia associated with spontaneous ventilation (nasal glasses with supplemental oxygen - Group 1) or treatment with general anesthesia under controlled mechanical ventilation (tidal volume from 6 to 8 ml / kg of the assumed weight and PEEP of 5 cmH2O - Group 2).

Sampling will be carried out for convenience, including patients routinely seen in the operating room of the hospitals involved and who meet the inclusion and exclusion criteria of this study. The allocation of patients will be performed through a table of random numbers generated prior to the beginning of the protocol. The process of randomization of patients in the groups will be carried out using random blocks. The method for blinding the study will be carried out using sealed envelopes and will include the blinding of the researchers, evaluators and those responsible for statistical analysis, but will not include the blinding of the attending physician and the patients.

The data will be stored in Excel and analyzed statistically using STATA 12.0 software. The statistical approach will be carried out through the "intention-to-treat" model. The assessment of ventilatory and hemodynamic parameters between the groups will be performed using ANOVA associated with Bonferroni for parametric data or the Kruskal-Wallis test associated with the Mann-Whitney test for nonparametric data. For categorical variables, we will use Fisher's exact test or Chi-square test. Repeated measures ANOVA will be used to assess outcomes between treatment groups over the follow-up period. In order to control important variables, such as surgical time, surgical complications, age, body mass index, and ASA classification (comorbidities), a statistical approach to assess confounding factors (linear regression model) will be performed after the period data collection. Results will be considered statistically significant when type I (P) error is less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ASA II to IV; age greater than 18 years; scheduled for arterial revascularization surgery on lower limbs.

Exclusion Criteria:

* Patients with a body mass index above 40 kg / m2 who underwent emergency surgery, with a history of pulmonary surgery, persistent hemodynamic instability in the preoperative period, history of asthma or chronic use of corticotherapy, or patients with history neuromuscular disorder. Patients with a history of use of anticoagulants or antiplatelet agents in the preoperative period who contraindicate the performance of spinal anesthesia will also be excluded from the study. In this study, only patients with peripheral vascular disease with critical and symptomatic ischemia in the lower limbs and scheduled to undergo elective arterial revascularization of the lower limbs will be included, and all patients with acute vascular obstruction or other associated vascular complications will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-02-28 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative pulmonary complications. | 7 days
  To evaluate the effects of spinal neuroaxial anesthesia under spontaneous ventilation (group 1) in relation to general anesthesia under mechanical ventilation (group 2) on the incidence of pulmonary complications (primary endpoint composed: mild respiratory failure / hypoxemia, severe respiratory failure, suspected pulmonary infection , atelectasis, acute lung injury, barotrauma, pulmonary infiltrate, pleural effusion, bronchospasm, cardiopulmonary edema, acute respiratory distress syndrome - ARDS) in the perioperative period of patients undergoing lower limb bypass surgery.

SECONDARY OUTCOMES:
Incidence of hemodynamic complications (secondary outcome consisting of distributive shock or persistent hypotension requiring use of vasoactive drugs) | 7 days
  To evaluate the effects of spinal neuroaxial anesthesia under spontaneous ventilation (group 1) in relation to general anesthesia under mechanical ventilation (group 2) on the incidence of hemodynamic complications (secondary outcome consisting of distributive shock or persistent hypotension requiring use of vasoactive drugs) in the perioperative period of patients undergoing lower limb bypass surgery.
Incidence of minor ventilatory complications related to the ventilation strategy (desaturation) in the intraoperative period. | 7 days
  To evaluate the effects of spinal neuroaxial anesthesia under spontaneous ventilation (group 1) in relation to general anesthesia under mechanical ventilation (group 2) on the incidence of minor ventilatory complications related to the ventilation strategy (desaturation) in the intraoperative period of patients undergoing lower limb bypass surgery.
Perioperative pulmonary, gasometric and inflammatory physiological parameters. | 7 days
  To evaluate the effects of spinal neuraxial anesthesia under spontaneous ventilation (group 1) in relation to general anesthesia under mechanical ventilation (group 2) on perioperative pulmonary, gasometric and inflammatory physiological parameters of patients undergoing lower limb bypass surgery.
Hemodynamic parameters in the perioperative period. | 7 days
  To evaluate the effects of spinal neuroaxial anesthesia under spontaneous ventilation (group 1) in relation to general anesthesia under mechanical ventilation (group 2) on hemodynamic parameters in the perioperative period of patients undergoing lower limb bypass surgery.
Incidence of various extrapulmonary complications, in-hospital mortality, length of stay in the post-recovery room -anesthetic, and length of hospital stay. | 7 days
  To evaluate the effects of spinal neuraxial anesthesia under spontaneous ventilation (group 1) in relation to general anesthesia under mechanical ventilation (group 2) on the incidence of various extrapulmonary complications (Annex 2), in-hospital mortality, length of stay in the post-recovery room -anesthetic, and length of hospital stay in patients undergoing lower limb bypass surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Andre P Schmidt, Principal Investigator — Hospital de Clinicas de Porto Alegre; Cristiano F Andrade, Study Chair — Hospital de Clinicas de Porto Alegre
Locations (1):
- Andre Prato Schmidt, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No